CLINICAL TRIAL: NCT01461525
Title: Comparison of Sphincter Preservation Surgery Versus Abdominoperineal Resection for Low Rectal Cancer: Prospective Clinical Trial
Brief Title: Comparison of Sphincter Preservation Surgery and Abdominoperineal Resection (APR): Prospective Clinical Trial
Acronym: ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other); National Cancer Center, Korea (Other Government); Seoul National University Boramae Hospital (Other); Hallym University Medical Center (Other); Daehang Hospital (Other)
Responsible Party: Principal Investigator, Sung-Bum Kang, Director of Colorectal Cancer Center, Principal Investigator, Professor, Seoul National University Bundang Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APR-SPS trial
Record Dates: First submitted 2011-10-20; First posted 2011-10-28 (Estimated); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Rectal Cancer
Keywords: Low Rectal Cancer; Sphincter preservation; Abdominoperineal resection; Quality of life; Sexual function; Urinary function; Oncologic outcome
MeSH Terms: conditions — Rectal Neoplasms | interventions — Proctectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sphincter preservation surgery (Experimental): Temporary ileostomy with anal sphincter preservation
  Interventions: Procedure: Sphincter preservation surgery
- Abdominoperineal Resection (Experimental): Permanent colostomy with total anal sphincter sacrifice
  Interventions: Procedure: Abdominoperineal resection

INTERVENTIONS:
Procedure: Abdominoperineal resection — After high ligation of IMA, TME with autonomic nerve preservation, proctectomy with sphincter sacrifice and permanent colostomy.
  Other Names: APR; Miles' operation
  Arms: Abdominoperineal Resection
Procedure: Sphincter preservation surgery — After high ligation of IMA, TME with autonomic nerve preservation, sphincter preservation and proctectomy with distal margin of more than 0.5cm in length and temporary ileostomy
  Other Names: SPS
  Arms: Sphincter preservation surgery

SUMMARY:
Sphincter preservation surgery in low rectal cancer has been increased due to better understanding of tumor biology and advances in surgical technology. Furthermore, a majority of patients prefer sphincter preservation rather than living with permanent colostomy. But it is not clear whether sphincter preservation is directly related with better quality of life. There have been many studies comparing sphincter preservation surgery and abdominoperineal resection in many aspects including oncologic and functional outcomes, and the quality of life. However, the conclusion remains controversial because of the different results between studies.

DETAILED DESCRIPTION:
This prospective study was designed to compare the quality of life after sphincter saving surgery and abdominoperineal resection. Because of ethical issues, it is difficult to conduct as a randomized trial. On the basis of tumor location, extent, and preoperative anal function, patient will be attributed to two different operative method groups. On the assumption that 10% of the patients are lost to follow-up at 1 year, at least 74 patients undergoing APR and 220 patients undergoing SPS will be recruited. The study will be continued until the target sample size will be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Low rectal cancer (5cm from anal verge by surgeon's digital rectal exam / rigid rectoscopy)
* Patient who understands and accepts to sign the informed consent form
* Confirmed preoperative colonoscopic biopsy (adenocarcinoma)
* Proper bone marrow function
* Proper renal function
* Proper liver function
* No severe comorbidity

Exclusion Criteria:

* Metastatic lesion detected in preoperative assessment
* Previous history of cancer disease. (except patients with skin cancer)
* Severe heart disease, congestive heart disease.
* Severe lung disease, respiratory failure.
* Mental illness.
* Invasion to prostate, bladder and combined resection needed (partial or radical.• Legally prohibited for clinical trial.
* Pregnancy or breast feeding.
* Previous disease or disability expected to influence the assessment of postoperative quality of life.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2011-10; Primary Completion 2019-08 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Quality of life outcome | 3 years
  Measured by EORTC-QLQ C30, CR38 questionnaires at preoperative(baseline)and postoperative(12,24,36 months).

SECONDARY OUTCOMES:
Oncologic outcomes | 5 years
  Oncologic outcomes (recurrence, survival)
Bladder function | 3 years
  Measured by IPSS questionnaire at preoperative(baseline)and postoperative(12,24,36 months).
Sexual function | 3 years
  Measured by FSFI,IIEF-5 questionnaires at preoperative(baseline)and postoperative(12,24,36 months).
Anal function | 3 years
  Only patients with sphincter preservation surgery, measured by manometry and MSKCC questionnaire at preoperative(baseline)and after ileostomy repair (12,24,36 months).

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Bum Kang, Ph. D., Principal Investigator — Seoul National University Bundang Hospital
Locations (6):
- South Korea (6):
  - Hallym University College of Medicine, Anyang-si, Gyeonggi-do
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul, Jongno-gu
  - Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul
  - Daehang Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang SB, Cho JR, Jeong SY, Oh JH, Ahn S, Choi S, Kim DW, Lee BH, Youk EG, Park SC, Heo SC, Lee DS, Ryoo SB, Park JW, Park HC, Lee SM, Kang SI, Kim MH, Oh HK, Shin R, Kim MJ, Lee KH, Kim YH, Kim JS, Lee KW, Lee HS, Kim HJ, Park YS, Sohn DK, Park KJ; Seoul Colorectal Research Group (SECOG). Quality of life after sphincter preservation surgery or abdominoperineal resection for low rectal cancer (ASPIRE): A long-term prospective, multicentre, cohort study. Lancet Reg Health West Pac. 2020 Dec 28;6:100087. doi: 10.1016/j.lanwpc.2020.100087. eCollection 2021 Jan. PMID 34327411